CLINICAL TRIAL: NCT04373291
Title: Using BCG Vaccine to Enhance Non-specific Protection of Health Care Workers During the COVID-19 Pandemic. A Randomized Controlled Multi-center Trial
Brief Title: Using BCG Vaccine to Protect Health Care Workers in the COVID-19 Pandemic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bandim Health Project (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: BCG-DENMARK-COVID; 2020-001888-90 (EudraCT Number)
Record Dates: First submitted 2020-05-01; First posted 2020-05-04 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Non-specific Effects of Vaccines; Morbidity; Absenteeism; Heterologous Immunity
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: A multi-center randomized placebo-controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to treatment. The physicians administering the BCG vaccine or placebo will not be blinded. In case of serious adverse events, the participant can be unblinded after consultation with the coordinating PI or sponsor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCG vaccine (Active Comparator): Participants that are randomized in the active arm will receive an adult 0.1 ml dose of BCG vaccine (BCG-Denmark, AJ Vaccines) in the skin covering the left upper deltoid muscle.
  Each 0.1 ml vaccine contains between 200000 to 800000 colony forming units of the live attenuated strain of Mycobacterium bovis (BCG), Danish strain 1331.
  Interventions: Biological: BCG-Denmark
- Control (Placebo Comparator): Placebo will be 0.1 ml sterile 0.9 % NaCl, which has a similar color as the resuspended BCG vaccine.
  Interventions: Biological: Saline

INTERVENTIONS:
Biological: BCG-Denmark — Participants randomized to receive BCG will receive one 0.1 ml dose of Mycobacterium bovis BCG live attenuated BCG-Denmark vaccine (AJ Vaccines, Copenhagen, Denmark) by intradermal injection in the left deltoid region.
  Arms: BCG vaccine
Biological: Saline — Participants randomized to the control group will receive one 0.1 ml dose sterile 0.9 % NaCl by intradermal injection in the left deltoid region.
  Arms: Control

SUMMARY:
Background: The COVID-19 pandemic challenges the available hospital capacity, and this will be augmented by absenteeism of healthcare workers (HCW). HCW are at high risk, currently HCW constitute 20% of all the COVID-19 cases in Denmark. Strategies to prevent absenteeism of HCW are urgently needed.

Bacille Calmette-Guérin (BCG) is a vaccine against tuberculosis, with protective non-specific effects against other infections; significant reductions in morbidity and mortality have been reported, and a plausible immunological mechanism has been identified.

We hypothesize that BCG vaccination can reduce HCW absenteeism during the COVID-19 pandemic.

Primary objective: To reduce absenteeism among HCW with direct patient contacts during the COVID-19 epidemic. Secondary objective: To reduce the number of HCW that are infected with SARS-CoV-2 during the COVID-19 epidemic and to reduce the number of hospital admissions amongst HCW with direct patient contacts during the COVID-19 epidemic.

Study design: A multi-center randomized placebo controlled trial. Study population: 1500 HCW with direct patient contacts; defined as nurses, physicians and other medical staff working at emergency rooms and wards where COVID-infected patients are treated.

Intervention: Participants will be randomized 1:1 to intradermal administration of a standard dose of BCG vaccine or placebo (saline).

Main study parameters/endpoints: Primary endpoint: Number of days of (unplanned) absenteeism for any reason. Secondary endpoints: Number of days of (unplanned) absenteeism because of documented COVID infection. Cumulative incidence of hospital admissions.

Risk for participants and impact: Based on previous experience and randomized controlled trials in adult and elderly individuals, the risks of BCG vaccination are considered low. The objective of this trial is to evaluate the potential beneficial effects of BCG vaccination through a lower work absenteeism rate of HCW and/or a mitigated clinical course of COVID infection.

DETAILED DESCRIPTION:
BACKGROUND Health-care workers face an elevated risk of exposure to - and infection with - SARS-CoV-2. It is imperative to ensure the safety, health and fitness of hospital personnel in order to safeguard continuous patient care. Strategies to prevent COVID-19 or to mitigate its clinical consequences are urgently needed.

Bacillus Calmette-Guérin (BCG) was developed as a vaccine against tuberculosis, but our group has shown that it can protect against death from other infections, it has what we have called non-specific effects (NSEs).[3] In clinical studies, BCG vaccination was associated with less child mortality, mainly as a result of reduced neonatal sepsis and respiratory infections. In a WHO-commissioned meta-analysis, BCG was associated with 42% (95%CI: 24-55%) lower child mortality.

NSEs of BCG are not limited to children. An Indonesian trial has shown that consecutive BCG vaccination for 3 months reduced the incidence of acute upper tract respiratory infections by 80% (95%CI=22-95%).

It has been recently demonstrated that the non-specific beneficial effects of BCG vaccination are due to epigenetic and metabolic reprogramming of innate immune cells, a process termed 'trained immunity'. E.g. among humans receiving yellow fever vaccine virus, those who had received BCG had - compared to placebo treated subjects - lower viral load, and improved anti-viral responses.

We hypothesize that BCG vaccination may induce (partial) protection against susceptibility to and/or severity of COVID-19. This study will evaluate the efficacy of BCG to improve the clinical course of COVID-19 and to prevent absenteeism.

Given the immediate threat of the COVID-19 epidemic the trial has been designed as a pragmatic study with a highly feasible primary endpoint, that can be continuously measured. We have therefore chosen unplanned absenteeism from work as primary outcome, in line with an ongoing clinical trial of BCG in the Netherlands.

OBJECTIVES Primary objective: To reduce absenteeism among HCW with direct patient contacts during the COVID-19 epidemic. Secondary objective: To reduce the number of HCW that are infected with SARS-CoV-2 during the COVID-19 epidemic and to reduce the number of hospital admissions amongst HCW with direct patient contacts during the COVID-19 epidemic.

HYPOTHESIS BCG vaccination of HCW will reduce absenteeism by 20% over a period of 6 months.

METHODS

Study design and follow-up:

A multi-center randomized placebo-controlled trial.

STUDY POPULATION As the COVID-19 epidemic has already started in Denmark, our intention is to start as soon as possible. Recruitment of study participants will take place at participating hospitals, at departments were COVID-19 patients are treated and, thus, the risk of exposure to SARS-CoV-2 is high.

Participating hospitals Hospital PI Odense University Hospital Isik Somuncu Johansen Sygehus Lillebælt, Kolding Poul-Erik Kofoed Hvidovre Hospital Thomas Lars Benfield Nordsjællands Hospital Ellen Løkkegaard Aarhus University Hospital Christian Wejse Herning Hospital Lars Skov Dalgaard Sygehus Sønderjylland Christian B. Mogensen

TREATMENT OF SUBJECTS Participants will be randomized 1:1 to receiving one intradermal BCG vaccine or placebo. Participants that are randomized in the active arm will receive a BCG vaccine (BCG-Denmark, AJ Vaccines). Placebo will be 0.1 ml sterile 0.9 % NaCl, which has a similar color as the resuspended BCG vaccine.

STUDY PROCEDURES Day 0: Participants fill in a short questionnaire regarding baseline characteristics. A blood sample will be drawn for subsequent testing for SARS-CoV-2 antibodies. Participants will be randomised to BCG or placebo in a 1:1 ratio. Randomisation will be done centrally using the REDCap tool with stratification per hospital and by age groups (+/- 45 years of age) in blocks of 8.

Participants will be blinded to treatment. The physicians administering the BCG vaccine or placebo will not be blinded. In case of serious adverse events, the participant can be unblinded after consultation with the coordinating PI or sponsor.

The end of the trial is defined as whichever comes latest: the last patient's last registration in the online data collection, or 180 days.

Day 0 till end of trial (weekly): Short electronic questionnaire regarding work absenteeism, symptoms and side effects through REDCap. In case a participant reports acute respiratory symptoms indicating COVID-19, he or she will be tested depending on test availability.

End of trial: Participants are asked to fill in a final questionnaire. A blood sample will be drawn for subsequent testing for SARS-CoV-2 antibodies.

STATISTICAL ANALYSIS All analyses will be performed from the intention-to-treat principle. The primary endpoint will be analysed as counts per week (i.e. multiple observations per subject) using a Bayesian negative binomial regression. Similar regression models will be used for secondary endpoints: Number of days of unplanned absenteeism because of documented COVID; number of days of self-reported fever. Documented COVID, death for any reason, death due to documented COVID, cumulative incidence of Intensive Care Admission for any reason, cumulative incidence of Intensive Care Admission due to documented COVID, cumulative incidence of Hospital Admission for any reason, cumulative incidence of Hospital Admission due to documented COVID will be analysed in Cox proportional hazards models.

Participants will be followed until a new vaccine is given (but data will also be analyzed after receipt of a new vaccine type, to study potential interactions).

When applicable (i.e. in the event that one or more participants have died during the follow-up period) a competing events analysis will be performed in addition.

Interim analysis Every month, an interim analysis will be conducted by the independent statistician of the trial. The parallel Dutch trial will enable combined analysis that will strengthen the conclusions and increase the power to analyse the secondary outcomes and more rare outcomes as intensive hospitalization.

ETHICAL CONSIDERATIONS The study has ben approved by the Ethics Committee and by the Danish Medicines Agency.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet the following criteria:

* Adult (≥18 years);
* Hospital personnel caring for patients with COVID-19.

Exclusion Criteria:

* Known allergy to (components of) the BCG vaccine or serious adverse events to prior BCG administration
* Known active or latent infection with Mycobacterium tuberculosis (M. tuberculosis) or other mycobacterial species
* Previous M. tuberculosis infection
* Previous confirmed COVID-19 infection
* Fever (>38 C) within the past 24 hours
* Suspicion of active viral or bacterial infection
* Pregnancy
* Severely immunocompromised subjects (This exclusion category comprises a) subjects with known infection by the human immunodeficiency virus (HIV-1); b) subjects with solid organ transplantation; c) subjects with bone marrow transplantation; d) subjects under chemotherapy; e) subjects with primary immunodeficiency; f) treatment with any anti-cytokine therapies. g) treatment with oral or intravenous steroids defined as daily doses of 10 mg prednisone or equivalent for longer than 3 months)
* Active solid or non-solid malignancy or lymphoma within the prior two years;
* Direct involvement in the design or the execution of the BCG-DENMARK-COVID study
* Employed to the hospital < 22 hours per week
* Not in possession of a smartphone/tablet.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1293 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of days of unplanned absenteeism for any reason | 6 months

SECONDARY OUTCOMES:
The cumulative incidence of documented COVID | 6 months
Cumulative incidence of all-cause and infectious hospital admissions, in particular respiratory infections | 6 months
The number of days of unplanned absenteeism, because of documented COVID | 6 months
Number of days of (unplanned) absenteeism due to infections | 6 months
Number of days of (unplanned) absenteeism due to respiratory infections | 6 months
The number of days of self-reported fever (≥38 °C) | 6 months
The number of days of absenteeism, because of imposed quarantine as a result of exposure to SARS-CoV-2 | 6 months
The number of days of unplanned absenteeism because of self-reported acute respiratory symptoms | 6 months
The number of days of absenteeism, because of imposed quarantine as a result of having acute respiratory symptoms, fever or documented SARS- CoV-2 infection | 6 months
The number of days of self-reported acute respiratory symptoms | 6 months
The cumulative incidence of death for any reason | 6 months
Cumulative incidence of infectious disease episodes, in particular respiratory infections | 6 months
The cumulative incidence of self-reported acute respiratory symptoms | 6 months
The cumulative incidence of death due to documented COVID | 6 months
The cumulative incidence of Intensive Care Admission for any reason | 6 months
The cumulative incidence of Intensive Care Admission due to documented COVID | 6 months
The cumulative incidence of Hospital Admission due to documented COVID | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Schaltz-Buchholzer, MD, Principal Investigator — Bandim Health Project, University of Southern Denmark; Anne Marie Rosendahl Madsen, MD, Principal Investigator — Bandim Health Project, University of Southern Denmark; Christine Stabell Benn, Professor, Study Chair — Bandim Health Project, University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Region Syddanmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable individual data can be shared on the basis of a data sharing proposal sent to cbenn@health.sdu.dk
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When follow-up has been completed and the dataset have been closed
Access Criteria: Non-identifiable individual data can be shared on the basis of a data sharing proposal sent to cbenn@health.sdu.dk

REFERENCES:
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Aaby P, Kollmann TR, Benn CS. Nonspecific effects of neonatal and infant vaccination: public-health, immunological and conceptual challenges. Nat Immunol. 2014 Oct;15(10):895-9. doi: 10.1038/ni.2961. PMID 25232810
- [Background] Biering-Sorensen S, Aaby P, Napirna BM, Roth A, Ravn H, Rodrigues A, Whittle H, Benn CS. Small randomized trial among low-birth-weight children receiving bacillus Calmette-Guerin vaccination at first health center contact. Pediatr Infect Dis J. 2012 Mar;31(3):306-8. doi: 10.1097/INF.0b013e3182458289. PMID 22189537
- [Background] Kristensen I, Aaby P, Jensen H. Routine vaccinations and child survival: follow up study in Guinea-Bissau, West Africa. BMJ. 2000 Dec 9;321(7274):1435-8. doi: 10.1136/bmj.321.7274.1435. PMID 11110734
- [Background] Aaby P, Roth A, Ravn H, Napirna BM, Rodrigues A, Lisse IM, Stensballe L, Diness BR, Lausch KR, Lund N, Biering-Sorensen S, Whittle H, Benn CS. Randomized trial of BCG vaccination at birth to low-birth-weight children: beneficial nonspecific effects in the neonatal period? J Infect Dis. 2011 Jul 15;204(2):245-52. doi: 10.1093/infdis/jir240. PMID 21673035
- [Background] Higgins JP, Soares-Weiser K, Lopez-Lopez JA, Kakourou A, Chaplin K, Christensen H, Martin NK, Sterne JA, Reingold AL. Association of BCG, DTP, and measles containing vaccines with childhood mortality: systematic review. BMJ. 2016 Oct 13;355:i5170. doi: 10.1136/bmj.i5170. PMID 27737834
- [Background] Wardhana, Datau EA, Sultana A, Mandang VV, Jim E. The efficacy of Bacillus Calmette-Guerin vaccinations for the prevention of acute upper respiratory tract infection in the elderly. Acta Med Indones. 2011 Jul;43(3):185-90. PMID 21979284
- [Background] Netea MG, Joosten LA, Latz E, Mills KH, Natoli G, Stunnenberg HG, O'Neill LA, Xavier RJ. Trained immunity: A program of innate immune memory in health and disease. Science. 2016 Apr 22;352(6284):aaf1098. doi: 10.1126/science.aaf1098. Epub 2016 Apr 21. PMID 27102489
- [Background] Spencer JC, Ganguly R, Waldman RH. Nonspecific protection of mice against influenza virus infection by local or systemic immunization with Bacille Calmette-Guerin. J Infect Dis. 1977 Aug;136(2):171-5. doi: 10.1093/infdis/136.2.171. PMID 894076
- [Background] Arts RJW, Moorlag SJCFM, Novakovic B, Li Y, Wang SY, Oosting M, Kumar V, Xavier RJ, Wijmenga C, Joosten LAB, Reusken CBEM, Benn CS, Aaby P, Koopmans MP, Stunnenberg HG, van Crevel R, Netea MG. BCG Vaccination Protects against Experimental Viral Infection in Humans through the Induction of Cytokines Associated with Trained Immunity. Cell Host Microbe. 2018 Jan 10;23(1):89-100.e5. doi: 10.1016/j.chom.2017.12.010. PMID 29324233
- [Background] Hatherill M, Geldenhuys H, Pienaar B, Suliman S, Chheng P, Debanne SM, Hoft DF, Boom WH, Hanekom WA, Johnson JL. Safety and reactogenicity of BCG revaccination with isoniazid pretreatment in TST positive adults. Vaccine. 2014 Jun 30;32(31):3982-8. doi: 10.1016/j.vaccine.2014.04.084. Epub 2014 May 9. PMID 24814553
- [Derived] Sovik WLM, Madsen AMR, Aaby P, Nielsen S, Benn CS, Schaltz-Buchholzer F. The association between BCG scars and self-reported chronic diseases: A cross-sectional observational study within an RCT of Danish health care workers. Vaccine. 2024 Mar 19;42(8):1966-1972. doi: 10.1016/j.vaccine.2024.02.049. Epub 2024 Feb 19. PMID 38378387
- [Derived] Madsen AMR, Schaltz-Buchholzer F, Benfield T, Bjerregaard-Andersen M, Dalgaard LS, Dam C, Ditlev SB, Faizi G, Johansen IS, Kofoed PE, Kristensen GS, Loekkegaard ECL, Mogensen CB, Mohamed L, Ostenfeld A, Oedegaard ES, Soerensen MK, Wejse C, Jensen AKG, Nielsen S, Krause TG, Netea MG, Aaby P, Benn CS. Using BCG vaccine to enhance non-specific protection of health care workers during the COVID-19 pandemic: A structured summary of a study protocol for a randomised controlled trial in Denmark. Trials. 2020 Sep 17;21(1):799. doi: 10.1186/s13063-020-04714-3. PMID 32943115
- See also: Novel Coronavirus (2019-nCoV) situation reports — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/situation-reports

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04373291/Prot_SAP_000.pdf